CLINICAL TRIAL: NCT06801626
Title: Novel Strategies for Reducing Burn Scar Itch
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-0180
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Burn Scar; Itch Scarring; Wound
Keywords: Itch; Burn; Diphenhydramine; Famotidine
MeSH Terms: conditions — Wounds and Injuries; Pruritus; Burns | interventions — Famotidine; Cromolyn Sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLUS Group (Experimental): Treatment with active H1 antihistamine and administered active H2 antihistamine and using cromolyn sodium PLUS (-PLUS active H1 antihistamine, plus active famotidine and active cromolyn sodium)
  Interventions: Combination Product: Famotidine and 4% topical cromolyn sodium
- Placebo Group (Placebo Comparator): Treatment with active H1 antihistamine plus administration of placebo famotidine and placebo cromolyn sodium.
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: Famotidine and 4% topical cromolyn sodium — Patients will be instructed to take a 20mg famotidine capsule twice daily, and to use the lotion (4% cromolyn sodium) twice daily.
  Arms: PLUS Group
Other: Placebo — Treatment with active H1 antihistamine plus administration of placebo famotidine and placebo cromolyn sodium.
  Arms: Placebo Group

SUMMARY:
The purpose of the study is to see whether using diphenhydramine (Benadryl), famotidine (Pepcid), and cromolyn sodium will decrease burn scar itch.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effect of a new approach to treating burn scar itch. In other patient populations experiencing itch, H2 antihistamines and/or topically applied cromolyn sodium have decreased itch. We believe that these medications will reduce itch from burn scars. To test this idea, the investigators will compare two methods of treating itch: 1) recommended oral diphenhydramine (Benadryl) with placebo capsule and placebo lotion and 2) recommended oral diphenhydramine (Benadryl) with administration of oral famotidine (Pepcid) and topically applied cromolyn sodium.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the inclusion criteria in order to be eligible to participate in the study.

* Participant has provided informed consent in a manner approved by the IRB and is willing and able to comply with the trial procedures.
* Adults: ≥18 to <80 years of age.
* Has an itchy burn scar.

Exclusion Criteria:

Participants meeting any of the exclusion criteria at baseline will be excluded from study participation.

* Failure to obtain consent or unable to return for follow up assessments.
* Patient is unable to follow the protocol required assessments.
* Member of a vulnerable class (e.g., prisoners, pregnant participant, etc.).
* Any medical condition that, in the opinion of the investigator or physician, would place the participant at increased risk for participation.
* Concurrent participation in another interventional clinical trial (to avoid confounding factors that may influence outcomes).
* History of prior non-compliance or the presence or history of psychiatric condition (including drug or alcohol addiction) that would, in the opinion of the investigator, make it difficult for the participant to comply with the study procedures or follow the investigators instructions.
* Age < 18 or ≥ 80 years.
* Taking one of the following medications: cefuroxime, dasatinib, delavirdine, neratinib, pazopanib, risedronate, or tizanidine.
* Has a pre-existing inflammatory or itchy skin disease.
* Is taking an H2 antihistamine for another indication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Itch Scale: Visual Analogue Scale Itch (VAS Itch) | baseline, weekly for 3 months, at 3 and 6 months (+/-15 days each timepoint) after start date
  Patients will score the severity of itch on the scale provided at study start, once weekly for 3 months, at the 3-month visit, and again at study end (6 months). Patients will rate their itch from 0 to 10. to measure the intensity of itchiness, where a patient marks a point on a line to indicate how severe their itch is, with zero representing "no itch" and 10 representing "worst imaginable itch." A higher score means a worse outcome.

SECONDARY OUTCOMES:
The Patient and Observer Scar Assessment Scale 3.0 | baseline, and at clinic visit approximately 3 months (±15 days) after study start
  The Patient and Observer Scar Assessment Scale (POSAS) is an established scale for assessing scars by both the patient and the observer. The overall opinion of the scar is reported on a scale of 1-10, with 1 being normal skin and 10 being the worst scar. (POSAS 3.0) will be filled out by the participant and a clinical observer to evaluate scar severity/quality.
Brisbane Burn Scar Impact Panel (BBSIP) | baseline, and at clinic visit approximately 3 months (±15 days) after study start
  BBSIP is a patient-reported outcome measure developed in consultation with burn survivors that takes approximately 10 minutes to complete; the specificity of this comprehensive questionnaire allows detection of changes in quality of life related to burn hypertrophic scar. Higher scores indicate a worse outcome.
PROMIS-29 | baseline, and at clinic visit approximately 3 months after study start (±15 days)
  This questionnaire will be administered to determine whether the effects of treatment impact quality of life as reported by the patient.
Pain scale: Visual Analog Scale for Pain (VAS Pain) | baseline, and at clinic visit approximately 3 months and 6 months after study start (±15 days)
  The VAS pain score is a simple and effective method used to measure patients' pain levels. This method is typically represented by a line ranging from 0 to 10, where 0 indicates no pain and 10 indicates the most severe pain. Patients are asked to mark a point on the line that corresponds to their level of pain.
Patient Global Impression of Change (PGIC) | baseline, and at clinic visit approximately 3 months after study start (±15 days)
  A global index that consists of 3 questions to which participants will rate the severity of 1) their PAH symptoms, 2) shortness of breath (SOB), and 3) fatigue. The minimum and maximum range of scores for each of the 3 individual questions was 1-5, with severity scale choices of 1=not present, 2=mild, 3=moderate, 4=severe, and 5=very severe. A higher score indicates a worse outcome.
Participants Activity with Fitbit | Month 1, 2, 3 (+15 days, each timepoint)
  Overall activity: To be captured via Fitbit on a daily basis to gauge overall activity. These data will be correlated with the itch and pain scales, as reduced activity is associated with pain and/or itch.

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Finnerty, PhD, Principal Investigator — University of Texas Medical Branch, Galveston
Locations (1):
- University of Texas Medical Branch, Galveston, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No